CLINICAL TRIAL: NCT03076684
Title: Gender Differences in the Metabolic Effects of Uric Acid
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Preliminary data collected and diets developed. Funding has ended and data used to support a larger application to test the hypothesis.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Elizabeth Parks, Professsor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2007093
Record Dates: First submitted 2017-03-01; First posted 2017-03-10 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — Allopurinol

STUDY DESIGN:
Intervention Model Description: There are three arms of this study: a diet-treated group, a drug-treated group and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- low-fructose diet (Experimental): Intervention: low-fructose Subjects will consume a four-month diet with the goal of reducing added sugar intake from ≥13% of energy to <5% of energy and keeping their weight stable.
  Interventions: Other: low-fructose diet
- allopurinol treatment (Experimental): Subjects participating in the allopurinol treatment arm will begin with an initial dose of drug of 100 mg/d p.o. daily for 2 wks. The dose is then slowly increased over the next 8 wks to achieve a serum uric acid concentration of 6 mg/dL (maximum allopurinol dose is 800 mg/d). Once uric acid reaches 6 mg/dL, the subject stays on this dose and is seen for the interim visit (4 months), at which time all procedures are repeated. After this, drug treatment continues for another 4 months and the subject returns for the final visit at 8 months. The same procedures performed at baseline are repeated at this time. The dose of allopurinol will be taken the morning of the final visit.
  Interventions: Drug: Allopurinol
- control arm (No Intervention): After completion of the baseline visit (procedures described above), subjects participating in the control arm are not seen again until the 4-month time point, when the same procedures performed at baseline are repeated, except for the MRI. Following this, they are seen again at 8-months, when all baseline procedures are repeated. Cardiac MRI and labeled water consumption occur at the baseline and final visits.

INTERVENTIONS:
Other: low-fructose diet — Subjects will consume a four-month diet with the goal of reducing added sugar intake from ≥13% of energy to <5% of energy and keeping their weight stable.
  Arms: low-fructose diet
Drug: Allopurinol — Subjects in the drug arm will take the drug allopurinol daily.
  Arms: allopurinol treatment

SUMMARY:
Increased stiffening of the heart and blood vessels is a predictor of heart disease. Stiffening has been found to be greater in women than men, which puts women with poor blood sugar control at a greater risk for heart disease than men. In women only, a molecule in the blood called uric acid can be elevated due to diets high in fructose consumption and it is thought to be a cause of heart and vessel stiffening. From previous research, we have found that restricting fructose in the diet lowers uric acid more in women than men. There is also a drug that can be used to lower uric acid. These findings suggest a potential approach to decrease vessel and heart stiffness in women. The present study will investigate fructose restriction in the diet and drug treatment to lower uric acid in the blood and its effects on heart disease risk in women compared to men.

DETAILED DESCRIPTION:
This project will use treatments from 4-8 months to lower uric acid in men and women. This study has three parts and each subject will participate in only one part. Tests that will be performed before and after treatment include measurements of body weight, blood pressure, blood vessel stiffness, heart stiffness, and blood lipids and glucose.

Part 1: Dietary treatment The overall goal of part 1 is to remove fructose and simple sugars from the diets of women and men at risk for future heart disease. Dietary fructose will be replaced with starchy foods to keep the research subjects' body weights stable. Subjects will be treated for 4 months and measurements of vascular and heart stiffness will be made before, during, and after treatment.

Part 2: Drug treatment The overall goal of part 2 is to treat women and men with mild elevations in blood uric acid for 8 months. The treatment will be allopurinol administration, ramping up the dose over a 2 month period to achieve a uric acid concentration of 6 mg/dL. Measurements of vascular and heart stiffness will be made before, during, and after.

Part 3: Control, no treatment These individuals will undergo the same baseline and follow-up tests as the other two parts but have no treatments.

Tests that will be completed before and after

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with characteristics of the metabolic syndrome.
2. 40-70 years of age
3. Overweight/obese subjects with BMI 25.1 - 40.0 kg/m2
4. Pre-diabetes defined as fasting glucose 100 - 125 mg/dL or 2h glucose 140 - 200 mg/dL
5. Habitual diets containing ≥ 13.0% of energy from added sugars
6. Serum uric acid ≥ 7.0 mg/dL for men and women

Exclusion Criteria:

1. Renal dysfunction (defined by glomerular filtration rate [GFR] <60), abnormal thyroid function or liver disease
2. Use of diuretics or azathioprine
3. Diabetes defined as fasting glucose ≥ 125 mg/dL or HbA1c ≥ 7%
4. Use of medications that interfere with lipid, protein, or carbohydrate metabolism, or occasional or regular tobacco use
5. Habitual diets with low content of added sugars (<5% of total energy)
6. History of gout , gouty arthritis, or uncontrolled hypertension
7. Pregnant
8. Vegetarian food restrictions (the diets consumed contain some meat, eggs and dairy)
9. Alcohol intake: females > 70 g/wk, males >140 g/wk
10. Inability to have an MRI

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
vessel stiffness | Change from baseline at 4 months
  blood vessel stiffness is measured non-invasively with pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Parks, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No